CLINICAL TRIAL: NCT06165874
Title: [68Ga]Ga-NOTA-RW102 PET Imaging in the Diagnosis of PD-L1-expressing Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-546
Record Dates: First submitted 2023-11-19; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Positron-Emission Tomography
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-small cell lung cancer (Experimental): Patients were recruited in the Department of Thoracic Surgery
  Interventions: Radiation: [68Ga]Ga-NOTA-RW102 PET Imaging

INTERVENTIONS:
Radiation: [68Ga]Ga-NOTA-RW102 PET Imaging — Intravenous injection of 1.8 MBq[0.05MCi]/kg of [68Ga]Ga-NOTA-RW102 in a single dose.

SUMMARY:
The aim of this study was to establish and optimize the imaging method of [68Ga]Ga-NOTA-RW102, as well as its physiological and pathological distribution characteristics, on the basis of which the diagnostic efficacy of the above imaging agent was evaluated in patients with non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD-L1-positive non-small cell lung cancer

  1. Age between 18 and 65 years old, gender is not limited.
  2. Patients with CT findings that can be occupied on the lung with a diameter greater than 1cm or more who have not undergone surgery.
  3. Lung cancer patients with a clinical diagnosis of positive PD-L1 expression;
  4. Written informed consent must be signed by the subject or his/her legal guardian or caregiver.
  5. Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Severe hepatic and renal insufficiency;
  2. Targeted therapy prior to radiotherapy or PET/CT scan. PD-L1 expression in existing lesions was assessed by immunohistochemistry using antibody clone 22C3. Renal function: serum creatinine less than or equal to the upper limit of the normal range;
  3. Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range.
  4. History of serious surgery in the last month.
  5. Those who have participated in other clinical trials during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Calculation and comparison of [68Ga]Ga-NOTA-RW102 radioactivity concentrations in focal and non-focal tissues | 90mins from time of injection
  Assessment of the efficacy of [68Ga]Ga-NOTA-RW102 in the diagnosis and differential diagnosis of non-small cell lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

REFERENCES:
- [Derived] Zhang Y, Cao M, Wu Y, Malih S, Xu D, Yang E, Younis MH, Lin W, Zhao H, Wang C, Liu Q, Engle JW, Rasaee MJ, Guan Y, Huang G, Liu J, Cai W, Xie F, Wei W. Preclinical development of novel PD-L1 tracers and first-in-human study of [68Ga]Ga-NOTA-RW102 in patients with lung cancers. J Immunother Cancer. 2024 Apr 5;12(4):e008794. doi: 10.1136/jitc-2024-008794. PMID 38580333